CLINICAL TRIAL: NCT01080378
Title: Developmental Pathways to Metabolic Diseases: To Investigate the Metabolic Effects of Birth Weight on Overweight and Obese Chinese Adults and Their Responses to Weight Loss Over 16 Weeks
Brief Title: Metabolic Effects of Birth Weight on Overweight and Obese Chinese Adults and Their Responses to Weight Loss
Acronym: SAMS-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Associate Professor Chong Yap Seng, National University of Singapore (NUHS)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DSRB C/09/604
Record Dates: First submitted 2010-02-28; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Healthy; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Higher Birth Weight (Other): 3447g to 3879g
  Interventions: Procedure: Dietary and Exercise Intervention
- Lower Birth Weight (Other): 2624g to 2964g
  Interventions: Procedure: Dietary and Exercise Intervention
- Normal Birth Weight (Other): 2965g to 3446g
  Interventions: Procedure: Dietary and Exercise Intervention

INTERVENTIONS:
Procedure: Dietary and Exercise Intervention — Participants will be enrolled into a 16 weeks weight loss programme that consists of (a) dietary interventions and (b) structured exercise sessions and (c) physical activity to achieve 7 - 10% decrease (more than 8 kg) in initial body weight in 16 weeks. They will be subjected to a caloric deficit of 40% of the subject's energy expenditure or 1000kcal, which ever it is higher. (allowance given for dietary control and physical activity).

SUMMARY:
The overall objective of this study is to investigate in depth the impact of birth weight on the nature of metabolic physiology, body composition and epigenetic differences of the different phenotypes of overweight and obese individuals who are otherwise overtly healthy. We also aim to determine the efficacy of a weight loss intervention on the above mentioned metabolic parameters in these individuals.

DETAILED DESCRIPTION:
There is an exponential rise in the prevalence of type 2 diabetes and obesity in Singapore coincident with rapid nutritional and socioeconomic transition. Differing birth weights, even in the normal ranges, predisposes individuals to the risk of type 2 diabetes and obesity. We aim to examine the causal pathways, developmental contribution and effects of a weight loss intervention to this differential by evaluating the hypothesis that genomic, birth weight, developmental, lifestyle and environmental factors contribute to the variation in phenotype observed in adults with obesity and metabolic syndrome.

Although there are many large studies that examined the effect of birth weight on the expression of obesity and the metabolic syndrome phenotype, most of these studies usually lack in-depth physiological and epigenetic/genomic studies due to their large sample sizes. We therefore aim to explore such detailed aspects of physiological and epigenetic/genomic profiles on smaller but statistically powered samples, focusing on evaluating body composition, nutritional and metabolic phenotype in relationship to epigenetic/genetic markers and developmental history. In addition, we examine the effects of a weight loss intervention on these parameters. This will assist in weighing the importance of developmental and genetic pathways in contributing to individual risk and the response and efficacy to an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent
2. Chinese males (aged 21-40)
3. Body mass index between 23-30 kg/m2
4. Total body fat content >24%
5. Sedentary adults < 1 episode of exercise > =30 min/week
6. Birth weight between 5-95% percentiles
7. Fasting glucose < 7 mmol/L
8. Normotensive, defined as BP < 140/90 mmHg and not on any antihypertensive agents

Exclusion Criteria:

1. Recent changes in weight of >5% over the past 6 months
2. Attempts to lose weight (weight not stable, exercises still changing and not in maintenance phase) over the past 6 months
3. Significant changes in diet over the past 6 months
4. Any use of weight reducing drugs in the past 6 months
5. Previous abdominal surgery (and bariatric surgery)
6. Any bleeding disorders which would preclude biopsies
7. Any use of investigational drugs in the past 6 months
8. Known allergy to insulin or local anaesthetics
9. Known allergy to milk or milk products (eg. Ensure, liquid meal)
10. Any serious illness requiring hospitalization or surgery in the past 6 months
11. Treatment with medications for hypertension, diabetes mellitus or dyslipidemia, epilepsy, ischemic heart disease
12. On anti-platelet agents, non-steroidal anti-inflammatory drugs (NSAIDs) or anticoagulants
13. Use of any prescription medication that cannot be safely discontinued within 14 days prior to study entry
14. Any use of corticosteroids in the past 6 months
15. Any other medications that could alter insulin resistance
16. History of surgery with metallic clips, staples or stents
17. Presence of cardiac pacemaker or other foreign body in any part of the body including tattoos
18. Mother no longer alive or unable to provide information on birth weight
19. Born premature (ie. not full term baby < 37 weeks of gestation age)

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-04

CONTACTS AND LOCATIONS:
Overall Officials: Yung Seng Lee, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - SGH Life Centre, Singapore